CLINICAL TRIAL: NCT00832780
Title: INST 0810: Phase II Study of Stereotactic Body Radiation Therapy Using Tomotherapy for Tumors of the Lung
Brief Title: Phase II Study of Stereotactic Body Radiation Therapy Using Tomotherapy for Tumors of the Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0810; NCI-2011-02943 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Solid Tumors
Keywords: Lung cancer; radiation therapy; SBRT; Stereotactic Body Radiation Therapy; Tomotherapy; other solid tumors
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation (SBRT) (Experimental): 60 Gy using 12 Gy per fraction over 5 fractions, to be given within 10 calendar days
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — A total of 60 Gy using 12 Gy per fraction over 5 fractions to be given within 10 calendar days. Each fraction of 12 Gy will be divided into 2 fractions of 6 Gy given in one day within 6 hours. Dose will be prescribed to the isodose line which covers at least 90% of the planning target volume. Dose homogeneity +/- 5%.
  Other Names: SBRT

SUMMARY:
The purpose of this study is to determine the response of lung tumors to radiation therapy. This study will be using a type of radiation therapy called tomotherapy. Tomotherapy is a relatively new kind of therapy which is able to focus a large amount of radiation to a small area with relatively less radiation to the surrounding non-cancerous part of the organ. This study is being done to find out if this technique is able to control the cancer better or not than the standard radiation and also to study its safety.

DETAILED DESCRIPTION:
The introduction of stereotactic body radiation therapy (SBRT) has allowed safe dose escalation in treatment regimens for cancer. Several studies have shown a radiation dose-response relationship for survival and local control for tumors of the lung, including cancer that originates in the lung (such as non-small cell lung cancer) as well as cancer that metastasizes to the lung.

The purpose of this study is to determine the response rate and toxicity of SBRT treatment of patients with lung tumors. This study will use a dose of 60 gray (Gy) in 5 fractions of 12 Gy. This provides a biological equivalent dose with alpha/beta ratio of 10 (BED10) of 132 Gy with the anticipation of achieving local control without increased toxicity. Previous studies have shown that the response rate with SBRT across multiple studies is approximately 50%, with an additional 25-40% of patients having stable disease. We hypothesize that this regimen will achieve a response rate of 70% with grade 3 toxicity of less than 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic confirmation of non small cell lung cancer or other solid primary tumor metastatic to lungs
2. Medically inoperable stage I or II non small cell lung cancer with negative lymph nodes or metastatic cancer to lung with less than or equal to 3 lesions
3. Age greater than or equal to 18 years old
4. Zubrod performance status less than or equal to 1
5. Negative pregnancy test for women of child bearing potential
6. Informed consent
7. Each lesion must be less than or equal to 5 cm in maximal diameter and multiple lesions must be less than or equal to 18 cm for the sum of the diameters in 3 dimensions. Example: 3 lesions each 2+2+2 cm have an aggregate diameter of 18 cm which is acceptable.
8. No prior radiation to lesions being treated
9. For metastatic disease to lung, primary tumor needs to be controlled (no evidence of progression on imaging for at least 2 months).

Exclusion Criteria:

1. Contraindications to radiation
2. Within or touching the zone of proximal bronchial tree defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi)
3. Pregnant or lactating females who chose to breast feed
4. Patients must have recovered from toxicity of prior therapy
5. Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
6. Cytologically positive pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Liem, M.D, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- Universtiy of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: University of New Mexico Cancer Center — http://cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiation (SBRT)
Started | 44
Completed | 19
Not Completed | 25
Not completed — Death | 16
Not completed — Lost to Follow-up | 4
Not completed — no reason given | 2
Not completed — other complicating condition | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- 60 Gy Using 12 Gy Per Fraction Over 5 Fractions: Radiation dose of 60 Gy administered in 5 fractions of 12 Gy each.
Arm/Group | 60 Gy Using 12 Gy Per Fraction Over 5 Fractions
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.42 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR):
Description: RR is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. RR is the sum of the percentage of patients who achieved a CR or PR. (RR = CR + PR)
Time Frame: 2 years
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 44
Number analyzed (tumors) | 50
tumors | 38

2. Secondary Outcome: Treatment Related Toxicity
Description: Toxicity will be evaluated per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Frequency and severity of adverse events will be tabulated and reported.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 44
participants
  cough | 4
  fatigue | 1
  chest wall pain | 7
  shortness of breath | 3
  wheeze | 1

3. Secondary Outcome: Overall Survival (OS)
Description: The time from treatment initiation to death by any cause
Time Frame: up to 67 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 44
months | 44 [24 to 67]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from treatment initiation to disease progression or death by any cause. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT): Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 44
Participants | 31

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. Complete response (CR): Disappearance of all evidence of target and non-target lesions. Partial response (P): >= 30% reduction from baseline in the sum of the longest diameter of all lesions. Stable Disease (SD): Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. CBR is the sum of the percentage of patients who achieve a CR, PR or SD (CBR = CR + PR + SD).
Time Frame: 2 years
Measure: Count of Units; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 44
Number analyzed (tumors) | 50
tumors | 41

ADVERSE EVENTS:
Time Frame: 6 years, 9 months
Arm/Group | Stereotactic Body Radiation (SBRT)
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 7/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation (SBRT) (N=44)
Agitation (Psychiatric disorders) | 1 (1)
Chest pain (Cardiac disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes